CLINICAL TRIAL: NCT07193394
Title: Tucatinib and Trastuzumab in HER3-mutant and HER2-not Amplified Metastatic Breast Cancer: a Proof of Concept Study (H3RAKLES)
Brief Title: Tucatinib and Trastuzumab in HER3-mutant and HER2-not Amplified Metastatic Breast Cancer
Acronym: H3RAKLES
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Pfizer (Industry); Eurofins (Industry); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IC 2024-01; 2024-519624-24-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-12; First posted 2025-09-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Breast Cancer ( HER2 Negative); Unresectable Breast Cancer
Keywords: Breast; Cancer; HER2; tucatinib; trastuzumab; HER3; metastatic; unresectable
MeSH Terms: conditions — Breast Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — tucatinib; Trastuzumab

STUDY DESIGN:
Intervention Model Description: The H3RAKLES single-arm phase II trial will evaluate the combination of tucatinib, a HER2 TKI, and trastuzumab, a HER2-directed antibody, with a Bayesian design in patients with a HER2-not amplified metastatic or unresectable breast cancer harboring an activating ERBB3 mutation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with tucatinib and trastuzumab combination (Experimental): Patients with HER2-not amplified metastatic or unresectable breast cancer harboring an activating ERBB3 mutation, treated with a combination of tucatinib and trastuzumab
  Interventions: Drug: Tucatinib (ONT-380); Drug: Trastuzumab (Herceptin)

INTERVENTIONS:
Drug: Tucatinib (ONT-380) — Patients with a HER2-not amplified metastatic or unresectable breast cancer harboring an activating ERBB3 mutation will receive experimental treatment with tucatinib and trastuzumab combination
Drug: Trastuzumab (Herceptin) — Patients with a HER2-not amplified metastatic or unresectable breast cancer harboring an activating ERBB3 mutation will receive experimental treatment with tucatinib and trastuzumab combination

SUMMARY:
The H3RAKLES trial would allow patients with a progressive metastatic breast cancer to have access to one more line of systemic therapy. Patients included in this trial will have already received at least two lines of chemotherapy (and potentially several lines of endocrine therapy for patients with a HR+ disease). In this setting, few treatments have demonstrated a clinically meaningful benefit, and any additional option is valuable. Furthermore, the pre-clinical and clinical rationale indicate a high probability of clinical benefit, as previously shown in Table 1, with all patients treated with trastuzumab and a TKI targeting HER2 displaying a response. Besides, with several years of hindsight for the combination of lapatinib, trastuzumab and capecitabine, we expect excellent tolerance with the same treatment without capecitabine.

The H3RAKLES single-arm phase II trial will evaluate the combination of tucatinib, a HER2 TKI, and trastuzumab, a HER2-directed antibody in patients with a HER2-not amplified metastatic or unresectable breast cancer harboring an activating ERBB3 mutation. To demonstrate the actionability of ERBB3 mutations, all patients will receive a combination of trastuzumab and tucatinib, in 3-weeks cycles.

DETAILED DESCRIPTION:
For breast cancers in which HER2 is not overexpressed, activating mutations in the ERBB3 gene, coding for the HER3 tyrosine kinase receptor, have an oncogenic role, and targeting them may offer new perspectives of treatment.

Pre-clinical data suggest that HER2 is essential for the pro-tumoral effect of HER3, which does not have a functional tyrosine kinase domain and requires heterodimerization with other members of the HER family of tyrosine kinase receptors for signaling. There is limited clinical evidence of the activity of drugs targeting HER2 in cancers harboring ERBB3 mutations, but few patients with breast cancer have been evaluated. Furthermore, the distribution of ERBB3 mutations seems to differ in breast carcinoma when compared to other cancer types. A few patients with a HER2 non-amplified metastatic breast cancer were treated at Institut Curie with the combination of a HER2-directed antibody and of a HER2 tyrosine kinase inhibitor (TKI) and all responded, warranting further explorations in this setting.

The H3RAKLES single-arm phase II trial will evaluate the combination of tucatinib, a HER2 TKI, and trastuzumab, a HER2-directed antibody, with a Bayesian design in patients with a HER2-not amplified metastatic or unresectable breast cancer harboring an activating ERBB3 mutation.

To demonstrate the actionability of ERBB3 mutations, all patients will receive a combination of trastuzumab and tucatinib, in 3-weeks cycles, until cancer progression, inacceptable toxicity or patient's withdrawal from the trial.

Tumor radiological assessments will be performed every 6 weeks during the 6 first months (first 8 cycles), then every 9 weeks until disease progression. In addition, Quality of Life will be evaluated throughout the treatment.

Blood samples (at baseline, cycles 1, 2 and 3, and at end of treatment) and tissue samples (at baseline and optionally at progression) will be collected as part as exploratory objective analyses on biomarkers (ctDNA monitoring and next-generation sequencing (NGS)).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Metastatic or unresectable breast cancer
* HER2-negative (defined as having an IHC 0+, IHC 1+, or IHC 2+ and ISH non-amplified, per ASCO/CAP guidelines) on last assessable tumor sample
* Having received ≥ 2 previous chemotherapy lines for advanced breast cancer: including at least one line of conjugated antibody, at the investigator's discretion or if a germinal BRCA mutation is present, a PARP inhibitor.
* Class IV or V somatic ERBB3 mutation as determined on a tumor sample obtained during the molecular screening step
* ECOG performance status ≤ 2 (Appendix A)
* Evaluable disease, per RECIST v1.1 inclusion criteria
* Left ventricular ejection fraction (LVEF) ≥50% as assessed by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA) documented within 4 weeks prior to first dose of study treatment
* Adequate organ function:

  1. Creatinine clearance ≥ 50 mL/min as calculated per institutional guidelines
  2. Total bilirubin ≤1.5 X upper limit of normal (ULN), except for patients with known Gilbert's disease, who may enroll if the conjugated bilirubin is ≤1.5 X ULN.
  3. Transaminases (aspartate aminotransferase and alanine aminotransferase) ≤ 2.5 X ULN (≤ 5 X ULN if the patient has liver metastases)
* Women of childbearing potential (WCBP) must have a negative serum pregnancy test < 7 days prior to first dose of treatment. A woman is considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. A postmenopausal state is defined as the absence of menses for 12 months without an alternative cause.
* WCBP (as defined above) and men with partners of childbearing potential must agree to use a highly effective birth control method during the study and for 3 months after completion of investigational treatment.
* Patients should be eligible for the treatment step according to the investigator's opinion.
* Patients must be covered by a health insurance plan.
* Patients able to provide signed informed consent.

Exclusion Criteria:

* Having received any prior treatment targeting HER2. Prior treatment with trastuzumab deruxtecan is allowed, per label, in patients with HER2-low metastatic breast cancer (IHC 1+ or 2+, ISH non-amplified)
* History of allergic reactions to trastuzumab or tucatinib or chemically similar drugs
* Patients who are pregnant, breastfeeding, or planning a pregnancy from time of informed consent until 7 months after the final dose of study drug
* Inability to swallow pills or having a significant gastro-intestinal disease or a history of surgery which would preclude the adequate oral absorption of medications
* Having used a strong CYP2C8 inhibitor within a duration of 5 half-lives prior to the first dose of study treatment, or have used a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment (see Appendix B and Appendix C)
* Treatment with any systemic anti-cancer therapy (including hormonal therapy), non-central nervous system (CNS) radiation, or experimental agent ≤ 3 weeks prior to the first dose of study treatment, except gonadotropin releasing hormone (GnRH) agonists
* Participation in another interventional clinical trial.
* Symptomatic and untreated brain metastases or brain metastases requiring urgent treatment, or brain metastases requiring a dose > 2 mg of dexamethasone (or equivalent)
* Whole brain radiotherapy < 21 days prior to first dose of treatment, stereotactic radiotherapy < 7 days prior to first dose of treatment
* Leptomeningeal metastases
* Major surgery (including surgery of brain metastases) < 21 days prior to first dose of treatment
* Evidence within 2 years of the start of study treatment of another malignancy that required systemic treatment
* Have known myocardial infarction or unstable angina within 24 weeks prior to first dose of study treatment
* Have clinically significant cardiopulmonary disease such as:

  * Ventricular arrhythmia requiring therapy,
  * Uncontrolled hypertension (defined as persistent systolic blood pressure >150 mmHg and/or diastolic blood pressure > 100 mm Hg on antihypertensive medications)
  * Any history of symptomatic congestive heart failure
  * Severe dyspnea at rest (CTCAE v5.0 Grade 3 or above) due to complications of advanced malignancy
  * Hypoxia requiring supplementary oxygen therapy except when oxygen therapy is needed only for obstructive sleep apnea
  * Presence of ≥ Grade 2 QTc prolongation on screening ECG
* Conditions potentially resulting in drug-induced prolongation of the QT interval or torsade de pointes:

  * Congenital or acquired long QT syndrome
  * Family history of sudden death
  * History of previous drug-induced QT prolongation
  * Current use of medications with known and accepted associated risk of QT prolongation (see row "Accepted Association" in Appendix D)
* Are known carriers of active Hepatitis B or Hepatitis C or have other known chronic liver disease
* Are known to be positive for human immunodeficiency virus (HIV)
* Altered mental status or psychiatric disorder that, in the opinion of the investigator, would preclude a valid patient informed consent.
* Patients who have difficulty undergoing trial procedures for geographic, social or psychological reasons
* Person deprived of liberty or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2028-12-07 (Estimated); Study Completion 2029-06-08 (Estimated)

PRIMARY OUTCOMES:
Clinical benefit rate (CBR) | 24 weeks
  Clinical benefit rate (CBR), defined as the proportion of patients who achieved a complete response (CR), a partial response (PR), or had stable disease (SD) for 24 weeks or more, according to the investigator-assessed RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 18 months
  Progression-free survival (PFS), defined as the time from inclusion to progression or death.
Overall survival (OS) | 18 months
  Overall survival (OS), defined as the time from inclusion to death by any cause.
Objective response rate (ORR) | 18 months
  Objective response rate, defined as the proportion of patients who achieved a CR or PR according to the investigator-assessed RECIST v1.1 criteria.
Safety of the trastuzumab/tucatinib combination | 18 months
  Adverse Events (AEs) and Serious Adverse Events (SAEs), per CTCAE v5.0, considered by the investigator as related to trastuzumab or tucatinib.

CONTACTS AND LOCATIONS:
Overall Officials: François-Clément Bidard, Prof., Principal Investigator — Institut Curie; Sandra BIDARD, Principal Investigator — Institut Curie
Locations (9):
- France (9):
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Chu Dupuytren- Limoges, Limoges
  - Institut Paoli-Calmettes, Marseille
  - Centre Antoine Lacassagne, Nice
  - CHU de Nîmes, Nîmes
  - Centre Eugène Marquis, Rennes
  - Institut Curie_ Site Saint-Cloud, Saint-Cloud
  - Institut Universitaire du Cancer de Toulouse (IUCT) - Oncopole Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
  IPD sharing Supporting Information: cases à cocher Study Protocol, Statistical Analysis Plan (SAP).
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).